CLINICAL TRIAL: NCT07400328
Title: A Single-Arm, Single-Center Exploratory Study of Amimestrocel Injection for the Prevention of Gastrointestinal Mucositis Induced by Conditioning Regimens Containing TBI and/or Melphalan
Brief Title: Amimestrocel Injection for Preventing Severe Oral Mucositis in HSCT Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SOOCHOW-WXJ-2025-1292
Record Dates: First submitted 2026-01-19; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Oral Mucositis; Stomatitis; Gastrointestinal Mucositis; Hematopoietic Stem Cell Transplantation
Keywords: Amimestrocel; Mesenchymal Stem Cells; Umbilical Cord; Mucositis Prevention; Total Body Irradiation; Melphalan; Conditioning Regimen; Allogeneic Transplantation; Single-Arm Trial
MeSH Terms: conditions — Stomatitis; Mucositis

STUDY DESIGN:
Intervention Model Description: This is a single-arm (single group assignment), open-label, exploratory study. All enrolled participants receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amimestrocel Injection (Experimental): All enrolled participants will receive a single, fixed-dose intravenous infusion of Amimestrocel injection (6.0×10⁷ cells in 12mL). The infusion is administered within 24 to 48 hours after the last dose of cyclophosphamide (part of the standard conditioning regimen) and before the infusion of hematopoietic stem cells (Day 0). All participants will also undergo standard myeloablative conditioning (containing TBI and/or melphalan), allogeneic hematopoietic stem cell transplantation, and institutional standard supportive care.
  Interventions: Biological: Amimestrocel injection

INTERVENTIONS:
Biological: Amimestrocel injection — Amimestrocel injection is an allogeneic (donor-derived), umbilical cord mesenchymal stem cell (UC-MSC) suspension for intravenous infusion. It is supplied as a cryopreserved cell suspension in a single-dose bag containing 6.0×10⁷ viable cells in 12 mL. For this study, a single bag is thawed and administered as a one-time intravenous infusion.
  Other Names: Ruibo Sheng

SUMMARY:
This study aims to see if a single intravenous infusion of a cell therapy called Amimestrocel injection can help prevent severe mouth sores (oral mucositis) in patients receiving a stem cell transplant.

Patients getting a stem cell transplant often receive strong chemotherapy (with radiation and/or a drug called melphalan) that can cause painful mouth and gut sores, making eating difficult and increasing infection risk. Amimestrocel injection is made from human umbilical cord cells that may help reduce inflammation and promote healing.

About 22 adult patients scheduled for this type of transplant at one hospital in China will receive the infusion 1-2 days before their stem cell transplant. Researchers will closely check for mouth sores, pain, and side effects for the first 28 days, and continue safety monitoring for 100 days.

The main goal is to see if the treatment lowers the rate of severe (Grade 3-4) mouth sores. The study will also track pain levels, need for pain medication, diarrhea, time for blood counts to recover, and overall safety.

DETAILED DESCRIPTION:
Background and Rationale:

Myeloablative conditioning regimens containing total body irradiation (TBI) and/or high-dose melphalan are standard prior to allogeneic hematopoietic stem cell transplantation (HSCT) but frequently cause severe gastrointestinal mucositis. This condition leads to significant morbidity, including pain, dysphagia, diarrhea, nutritional impairment, infection risk, prolonged hospitalization, and increased costs. Effective preventive strategies are limited. Mesenchymal stem cells (MSCs) have demonstrated immunomodulatory and tissue-repair properties via paracrine secretion of anti-inflammatory and growth factors, showing potential in mitigating mucosal injury in preclinical and early clinical contexts.

Study Design:

This is a single-arm, single-center, open-label, exploratory interventional study. It will enroll approximately 22 subjects to preliminarily evaluate the efficacy and safety of prophylactic Amimestrocel infusion.

Intervention:

Eligible patients will receive a single, fixed-dose intravenous infusion of Amimestrocel injection (6.0×10⁷ cells in 150 mL) within 24 to 48 hours after the last dose of cyclophosphamide (part of the standard conditioning regimen) and before the infusion of hematopoietic stem cells (Day 0).

Study Population:

Adults aged 18-65 years planned for myeloablative allogeneic HSCT with a TBI and/or melphalan-containing conditioning regimen, with adequate organ function and ECOG status 0-1. Key exclusions include active uncontrolled infection, allergy to MSCs, prior cell therapy, and pregnancy.

Endpoints and Assessments:

Primary Endpoint: Incidence of Grade 3-4 oral mucositis (assessed daily by WHO/NCI-CTCAE criteria) within 28 days post-transplant (Day 0 to +28).

Secondary Endpoints: Duration/severity of oral and gastrointestinal mucositis; oral pain (Numerical Rating Scale); opioid use; time to neutrophil engraftment (ANC ≥0.5×10⁹/L); incidence of adverse events and serious adverse events (monitored until Day +100).

Sample Size Justification:

The sample size of 22 is derived from an assumption of reducing the historical incidence of severe oral mucositis (71% based on literature) to 41% (30% absolute reduction), with 80% power and a two-sided alpha of 0.05, accounting for a 10% dropout rate.

Study Procedures Overview:

The process includes a screening period (Day -14 to -7), the investigational product infusion, an intensive observation phase (Day 0 to +28) with daily mucositis and pain assessments, and a safety follow-up phase until Day +100 for AE/SAE monitoring, GVHD, and survival status.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years.
2. Planned to undergo myeloablative allogeneic hematopoietic stem cell transplantation.
3. The conditioning regimen must contain total body irradiation (TBI) and/or melphalan.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Adequate organ function defined as:Left ventricular ejection fraction (LVEF) ≥ 50%.Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN).Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min.
6. Voluntarily signs the informed consent form.

Exclusion Criteria:

1. History of allergy to mesenchymal stem cells or any component of the Amimestrocel injection preparation.
2. Presence of active, uncontrolled bacterial, fungal, or viral infection.
3. History of other malignancies within the past 5 years, except for cured carcinoma in situ or basal cell skin cancer.
4. Pregnant or lactating women, or those planning pregnancy during the study period.
5. Previous receipt of any cell therapy product.
6. Severe psychiatric disorder or cognitive impairment that would limit the ability to provide informed consent or comply with study procedures.
7. Any condition that, in the investigator's judgment, makes the subject unsuitable for study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3-4 Oral Mucositis within 28 Days Post-Transplant | From stem cell infusion (Day 0) up to Day 28 post-transplant
  The proportion of subjects who develop severe (Grade 3 or 4) oral mucositis from the transplant day (Day 0) up to Day 28 post-transplant. The severity of oral mucositis is assessed daily and the highest grade recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Maximum Severity Grade of Oral Mucositis | From Day 0 up to Day 28 post-transplant.
  The highest severity grade of oral mucositis experienced by the subject from Day 0 to Day 28 post-transplant. Grading is based on the NCI CTCAE v5.0 criteria (Grades 1-5). Results are described as the number and percentage of patients in each grade.
Duration of Oral Mucositis | From Day 0 up to Day 28 post-transplant.
  The number of days from the first date of onset of ≥ Grade 2 oral mucositis to the first date it resolves to ≤ Grade 1. For subjects who do not develop ≥ Grade 2 mucositis or whose condition does not resolve to ≤ Grade 1 within 28 days, the duration will be censored. Results are described as median and interquartile range.
Maximum Severity Grade of Diarrhea | From Day 0 up to Day 28 post-transplant.
  The highest severity grade of non-infectious diarrhea experienced by the subject from Day 0 to Day 28 post-transplant. Grading is based on the NCI CTCAE v5.0 criteria (Grades 1-5). Results are described as the number and percentage of patients in each grade.
Total Duration of ≥ Grade 2 Diarrhea | From Day 0 up to Day 28 post-transplant.
  The sum total of days the subject experiences non-infectious diarrhea of severity ≥ Grade 2 from Day 0 to Day 28 post-transplant. Results are described as median and interquartile range.
Peak Oral Pain Score | The highest score recorded in the subject's daily self-assessed oral pain Numerical Rating Scale (NRS, 0-10) from Day 0 to Day 28 post-transplant. Results are described as median and interquartile range.
  The highest score recorded in the subject's daily self-assessed oral pain Numerical Rating Scale (NRS, 0-10) from Day 0 to Day 28 post-transplant. Results are described as median and interquartile range.
Total Opioid Use from Day 0 to Day 28 Post-Transplant | From Day 0 up to Day 28 post-transplant.
  The total consumption of opioids for controlling oral mucositis-related pain from Day 0 to Day 28 post-transplant, converted to oral morphine milligram equivalents (MME). Results are described as median and interquartile range.
Time to Neutrophil Engraftment | From Day 0 up to Day 60 post-transplant.
  The number of days from Day 0 to the first of three consecutive days with an absolute neutrophil count (ANC) ≥ 0.5 × 10⁹/L. Estimated using the Kaplan-Meier method.
Incidence of Any Adverse Event (AE) within 100 Days Post-Transplant | From after investigational product infusion up to Day 100 post-transplant.
  The proportion of subjects who experience any grade of adverse event (AE) from after the investigational product infusion up to Day 100 post-transplant. The severity and relationship to the investigational product are assessed according to NCI CTCAE v5.0 criteria and protocol specifications.
Incidence of Serious Adverse Events (SAEs) within 100 Days Post-Transplant | From after investigational product infusion up to Day 100 post-transplant.
  The proportion of subjects who experience any serious adverse event (SAE) from after the investigational product infusion up to Day 100 post-transplant. SAE definition follows ICH-GCP guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: xiaojin Wu, Principal Investigator, Principal Investigator — The First Affiliated Hospital of Soochow University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nakagaki M, Kennedy GA, Gavin NC, Clavarino A, Whitfield K. The incidence of severe oral mucositis in patients undergoing different conditioning regimens in haematopoietic stem cell transplantation. Support Care Cancer. 2022 Nov;30(11):9141-9149. doi: 10.1007/s00520-022-07328-4. Epub 2022 Aug 26. PMID 36008731
- [Background] Kebriaei P, Hayes J, Daly A, Uberti J, Marks DI, Soiffer R, Waller EK, Burke E, Skerrett D, Shpall E, Martin PJ. A Phase 3 Randomized Study of Remestemcel-L versus Placebo Added to Second-Line Therapy in Patients with Steroid-Refractory Acute Graft-versus-Host Disease. Biol Blood Marrow Transplant. 2020 May;26(5):835-844. doi: 10.1016/j.bbmt.2019.08.029. Epub 2019 Sep 7. PMID 31505228
- [Result] Lv K, Gao B, Ye W, Shen C, Chen T, Wang C, Yao H. Promotion of Epithelial Healing in Oral Mucositis by hESC-derived Mesenchymal Stem Cells via the PI3K/AKT Pathway. Curr Stem Cell Res Ther. 2025;20(7):810-823. doi: 10.2174/011574888X338333241010104024. PMID 41147081
- [Result] Le Blanc K, Frassoni F, Ball L, Locatelli F, Roelofs H, Lewis I, Lanino E, Sundberg B, Bernardo ME, Remberger M, Dini G, Egeler RM, Bacigalupo A, Fibbe W, Ringden O; Developmental Committee of the European Group for Blood and Marrow Transplantation. Mesenchymal stem cells for treatment of steroid-resistant, severe, acute graft-versus-host disease: a phase II study. Lancet. 2008 May 10;371(9624):1579-86. doi: 10.1016/S0140-6736(08)60690-X. PMID 18468541
- [Result] Sonis ST. The pathobiology of mucositis. Nat Rev Cancer. 2004 Apr;4(4):277-84. doi: 10.1038/nrc1318. No abstract available. PMID 15057287

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT07400328/Prot_SAP_000.pdf